CLINICAL TRIAL: NCT04739540
Title: Food Insecurity Screening and Intervention: From Hospital to Home
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michelle Lopez, Assistance Professor Pediatrics- Hospital Medicine, Baylor College of Medicine
Other Study IDs: H-48108
Record Dates: First submitted 2021-01-13; First posted 2021-02-04 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Food Insecurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Food insecurity (FI), limited access to food due to a lack of money or other resources, affected an estimated 14% households with children in the US in 2018. Multiple national organizations, including the American Academy of Pediatrics (AAP), have identified adverse childhood outcomes that are strongly correlated with FI, and the AAP recommends that physicians universally screen for and address FI, but screening for FI has primarily been addressed in the outpatient setting. Recent data demonstrates rising FI needs related to COVID-19 pandemic. There is limited information regarding screening and interventions for inpatient FI, defined as the inability to obtain adequate food during hospitalization. Previous work performed a cross-sectional study of 200 caregivers of hospitalized children in Chicago, Illinois, estimated the prevalence of inpatient FI to be 32%. Locally, work by Drs. Alice Lee, Lopez, and Bocchini identified hospital food insecurity (FI) in 43% of the caregivers of hospitalized children (Lee, Alice, et al. "Food Insecurity in the Caregivers of Hospitalized Pediatric Patients." Pediatrics 2018: 481-481.) . The investigators also found a strong association between inpatient and household food insecurity. Hospital food insecurity has a profound effect on caregiver's ability to participate in caring for their children during the hospitalization. Currently, there is not a valid screening tool to address inpatient food insecurity and there is a paucity of data on the effects of FI interventions implemented in the hospital setting. Additionally, there is new data from the COVID Impact Survey and The Hamilton Project/Future of the Middle Class Initiative Survey of Mothers with Young Children demonstrating that FI prevalence has more than doubled in household with children.

DETAILED DESCRIPTION:
Screening / Enrollment: At enrollment the research coordinator will create daily epic report list, maintain notes on eligible subjects obtain informed consent, verify eligibility, have caregiver complete demographics questionnaire in REDCap, and have caregiver complete food insecurity survey in REDCap. Research coordinator will notify investigator of + FI screen based on score of 3 or higher for household or inpatient tallied in REDCap. Research coordinator to activate the Admission/Discharge/Transfers (ADT) notice in Epic and link the subjects child in order to be notified when subjects child is discharged. The investigator will verify the score for food insecurity positive caregivers and the investigator will order the caregiver tray or notify the RC that the RC can order the caregiver tray for FI positive caregivers in Epic. The RC will complete a brief study note in Epic to state the caregiver was enrolled in the study. The investigator will complete the referral to Texas Children's Hospital food bank representative. Parents will receive handouts on caregiver tray, guest tray, hospital food resources, and the FIRST link program with the Houston food bank phone number (found in attachments).

All study procedures will be completed after informed consent is obtained. If a caregiver declines to participate in the study or screens negative for FI, they will still have the option to meet with with social work who is able to provide FI resources including caregiver trays, food bank referrals, educational materials, and gift cards depending on the social workers assessment.

Follow up: Research coordinator will complete the follow up survey with caregiver 2 weeks after discharge. Subjects should be called daily (Mon-Friday) due to short window for follow up (2 weeks after discharge + 7 days). The RC will attempt to contact the subject at least three times by phone and one time by email in an attempt to complete the follow-up study visit and will notify PI about the non-availability of the subject to complete it. Responses will be entered into RedCAP by the RC if the survey is conducted by phone.

In order to objective data on whether the inpatient intervention was utilized by families the investigators will request a caregiver tray report from Morrison's food vendor company for the caregiver trays. The report request will include all caregiver trays ordered for West Tower 15, 14, and 12 floors: -Person who placed the order -Patient room number -Number of trays ordered -Time and date trays ordered -Meal ordered

Study staff will periodically run EPIC reports to determine the number of caregiver trays ordered for the study. This report will be used to reimburse social work for the cost of the food trays.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver (parent or legal representative who self-identifies as a primary caregiver) of a child admitted to West Tower acute care floors 12th, 14th and 15th at Texas Childrens Hospital Medical Center Campus. Study procedures will not involve the child directly.
* Age > 18 years old.
* English or Spanish speaking
* Hospital day 3 or greater

Exclusion Criteria:

* Caregiver at bedside is not the primary caregiver of the child as confirmed at time of informed consent.
* Previous enrollment on this study.
* Adolescent and Rehabilitation designated beds on 14th and 12th floors respectively.
* Confirmed COVID-19 positive patients under enhanced respiratory precautions because the caregivers for these patients are receiving food trays provided to them by the unit. (Caregivers of patients who are under investigation for COVID will not be enrolled until after the test is negative.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary caregiver that is defined as the parent or legal representative who self identifies as a primary caregiver for the child.
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of Food Insecurity | Up to 3 weeks
  The primary outcome is prevalence of food insecurity.

SECONDARY OUTCOMES:
Percentage of Patients Enrolled in Food Insecurity | 6 months
  Secondary outcomes are percentage of patients completing Houston Food Bank referral, and the percentage of patients who enroll in one or more food resource.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lopez, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States